CLINICAL TRIAL: NCT02444156
Title: Indoor Rowing in Adults With Impaired Glucose Regulation: a Pilot Study
Brief Title: Rowing Away From Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: Medtronic (Industry); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0492
Record Dates: First submitted 2015-05-07; First posted 2015-05-14 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus, Type 2; Glucose Intolerance; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise training (Experimental): All participants will receive usual care, including standard advice about diet and physical activity. In addition to usual care, participants will be asked to take part in a 12-week exercise programme. Participants will use an indoor rower (Concept 2, Model E) three times per week at Leicester Diabetes Centre. Each session will be supervised and the investigators will liaise with the participants to arrange convenient times to exercise, including mornings and evenings. The supervisors will teach the participants how to row correctly.
  Interventions: Other: Indoor rowing

INTERVENTIONS:
Other: Indoor rowing

SUMMARY:
Primary research question: What is the effect of indoor rowing, under the ideal circumstances of a laboratory setting, on glucose control in adults with impaired glucose control?

Secondary research question: Is it possible to develop a full-scale study of the benefits of indoor rowing under the usual circumstances of a community setting?

Why? It is good practice to conduct a small pilot study before embarking on an expensive full-scale study.

What? Around 150 minutes of aerobic exercise and around 150 minutes of resistance exercise per week are necessary to meet prevailing recommendations for adults with impaired glucose control. Around 120 minutes of indoor rowing per week might be a less time-consuming alternative to prevailing recommendations because indoor rowing involves a combination of aerobic and resistance exercise.

Who? Twenty men and postmenopausal women aged 45-65 years with impaired glucose regulation, such as those with type 2 diabetes. Eligible volunteers will not have smoked in the last year, will not have exercised regularly in the last six months, and will not be taking any form of diabetes medication other than metformin. Eligible volunteers will have stable weight and a body mass index of 25-40.

Where and how? Before and after the exercise intervention, glucose control (postprandial blood glucose concentrations) will be assessed at Leicester Diabetes Centre and cardiac function (MRI) will be assessed at Glenfield Hospital. During the exercise intervention, participants will use an indoor rower three times per week for 12 weeks at Leicester Diabetes Centre. Participants will be taught how to row correctly and the duration and intensity will gradually increase. In order to inform the design of a full-scale trial, recruitment rate will be assessed, adherence will be monitored, and a third party will interview participants to find out if the intervention and assessments are feasible and acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Participant is willing to allow their general practitioner to be informed of any incidental findings.
* Eligible men will be 45 to 65 years of age.
* Eligible women will be 45 to 65 years of age and will be postmenopausal, defined as no menstrual period in the last 12 months.
* Body mass index of 25 to 40 kg·m-2.
* Stable weight, defined as self-reported weight change of less than 5 kg in the last six months.
* Impaired glucose regulation, defined as impaired fasting glucose (fasting plasma glucose of 5.6 to 6.9 mmol·l-1), or impaired glucose tolerance (two-hour plasma glucose in the 75-g oral glucose tolerance test of 7.8 to 11.0 mmol·l-1), or haemoglobin A1C of 6.0% or greater, or type 2 diabetes (fasting plasma glucose of 7.0 mmol·l-1 or greater on two occasions).
* Volunteers with type 2 diabetes will either be treatment naïve or will have been taking a stable dose of metformin for at least four weeks prior to study entry.
* White European ethnicity. There are ethnic differences in cardiovascular disease risk and prevailing definitions of dyslipidaemia, insulin resistance and diabetes cannot account for these differences (Forouhi et al., Diabetologia, 2006, 49, 2580-8; Tillin et al., Journal of the American College of Cardiology, 2013, 61, 1777-86). Therefore, in order to make valid inferences, the investigators will only include white Europeans on this occasion.
* Little or no participation in exercise: eligible volunteers will not have been exercising two or more times per week for 20 minutes or longer for the last six months.

Exclusion Criteria:

* Volunteers with type 2 diabetes will be excluded if they are taking any form of diabetes medication other than metformin.
* Known cardiovascular disease.
* Symptoms of angina.
* Resting systole blood pressure ≥180 mm Hg or diastolic blood pressure ≥110 mm Hg.
* Statin use.
* Beta-blocker use.
* Verapamil use.
* Hormone replacement therapy.
* Any smoking in the last year.
* Any absolute contraindication to exercise testing.
* Abnormal exercise test.
* Inability to undertake an exercise programme for any reason.
* Participation in a research study involving an investigational produce in the past 12 weeks.
* Female volunteers who are pregnant, lactating or planning pregnancy during the course of the study. Pregnancy will be discussed during the consent procedure and the investigators will provide those in any doubt with a pregnancy test kit.
* Chronic kidney disease (EGFR of ≤30).
* Any metal implants.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in Glucose control | Changes from baseline (week 0) to post intervention (week 0 versus week 13 and week 0 versus week 14)
  Glucose control is indicated by postprandial glucose concentration, which will be assessed using a standardized meal test.
Change in Cardiac function | Changes from baseline (week 0) to post intervention (week 13)
  Cardiac function is indicated by diastolic strain rate, which will be assessed using magnetic resonance imaging.

SECONDARY OUTCOMES:
Recruitment rate | Response rate to up to seven months of recruitment
  Participants will be recruited via general practice databases and the investigators will calculate the proportion of eligible-and-invited individuals who agree to take part in the study.
Feasibility and acceptability as assessed by Semi-structured interviews | Semi-structured interviews will be conducted during (week 5 or 6) and after (week 14) the intervention
  The interview during the intervention will focus on recruitment literature, screening procedures, baseline assessments, and first impressions of indoor rowing. The interview after the intervention will focus on participants' experiences of indoor rowing, including their likes, dislikes and suggestions. Each interview will last around 30 to 60 minutes and will be led by an independent researcher not involved in the day-to-day conduct of the study. Some questions and topics will be predetermined, but conversations will be allowed to flow freely and change according to the interviewer's discretion.
Change in Sample size in a full-scale trial | Changes from baseline (week 0) to post intervention (week 13)
  Haemoglobin A1C is a longer-term marker of glucose control and may be an appropriate outcome for a full-scale trial. The investigators wish to use the sample standard deviation from this pilot study in haemoglobin A1C (and, possibly, other variables) to estimate the population standard deviation and, thus, the power of a full-scale trial.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Davies, MD, Principal Investigator — University of Leicester
Locations (1):
- Leicester Diabetes Centre, Leicester, United Kingdom